CLINICAL TRIAL: NCT04180904
Title: Diet Interventions in Psoriatic Arthritis
Acronym: DIPSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Women's College Hospital (Other); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 834176
Record Dates: First submitted 2019-11-14; First posted 2019-11-29 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Psoriatic Arthritis
Keywords: PsA (Psoriatic Arthritis), Diet, Food, Nutrition
MeSH Terms: conditions — Arthritis, Psoriatic; Salivary Gland Adenoma, Pleomorphic

STUDY DESIGN:
Intervention Model Description: In this randomized controlled pilot trial, we will test different diets to determine the impact on disease outcomes among patients with psoriatic arthritis. This is a 24-week trial that will enroll 90 patients with active psoriatic arthritis despite stable therapy among three sites in the US and Canada. Dietary interventions will be enhanced with gamification, including feedback and competition. Biomarker samples including blood, urine and stool specimens will be collected and banked for exploratory analyses.
Who Masked: Outcomes Assessor
Masking Description: In a study assessing dietary behavioral interventions, absolute blinding of the participants is not possible because of obvious differences between intervention diets. However, we will avoid naming the allocated dietary intervention and withhold information about our research hypothesis from the patients. Participants in the control group will receive the same schedule of visits and patient reported outcomes. The study rheumatologists (outcome assessors) will be blinded to the allocated group and the participants will be asked to avoid discussing the details of their diet with them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diet 1 (Active Comparator): Diet 1 will focus on the dietary pattern and monitor types of foods, supplementary nutrition, and provide nutritional support with a dietitian.
  Interventions: Other: Diet 1
- Diet 2 (Active Comparator): Diet 2 will focus on the dietary pattern and monitor the amount of food, complimentary nutrition, and nutritional support with a dietitian.
  Interventions: Other: Diet 2
- Diet 3 (No Intervention): Diet 3 will focus on healthy dietary patterns and provide nutritional support with a dietitian.

INTERVENTIONS:
Other: Diet 1 — Diet 1 will focus on which foods are eaten and the impact on disease outcomes.
  Arms: Diet 1
Other: Diet 2 — This diet will limit the amount of food energy consumed each day and the impact on disease outcomes. This will be determined by factors including the subject's demographics (age, sex, weight, height).
  Arms: Diet 2

SUMMARY:
The purpose of this study is to learn whether changing diet impacts psoriatic arthritis (PsA).

DETAILED DESCRIPTION:
The study asks if dietary change and nutritional support improves disease activity and if patients are better able to improve or sustain progress with additional incentives. The study will use an online program to communicate with participants through text and online surveys. This 24-week trial will enroll 90 patients in the US and Canada with New York University as a back-up site.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Required Rheumatologist-confirmed diagnosis of PsA fulfilling Classification of Psoriatic Arthritis Criteria (CASPAR)
* Willing to alter diet and participate for 24 weeks
* Able to attend follow-up visits
* Body mass index (BMI) > 25 and <40
* No history of eating disorders such as anorexia or bulimia
* Disease Activity in Psoriatic Arthritis Assessment (DAPSA) > 10
* Stable treatment for PsA for ≥3 months prior to enrollment (patients may be on any disease modifying anti-rheumatic drugs (DMARDs) or they can be free of systemic medications
* Owns and uses an iPhone or Android smart phone, or is willing to use a device provided by the study team

Exclusion Criteria:

* Inability to provide informed consent
* Plan to change systemic treatment for psoriasis or PsA in the next 4-8 weeks
* Use of systemic corticosteroids
* All persons who would be placed at an increased risk including any medical condition that will impair the ability of the person to participate in a nutritional intervention study (e.g. insulin dependent diabetes, use of coumadin, advanced malignancy, inflammatory bowel disease, dementia)
* History of food allergy to any of the components of olive oil or nuts
* Inability to read and write in English
* Unwillingness to change dietary habits
* Known pregnancy (pregnancy testing will be performed for women of childbearing age; weight changes will not accurately reflect the changes we would anticipate in pregnant patients and weight loss may be detrimental to maternal and/or fetal outcomes).
* Participation in another physical activity study and/or diet trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Change in Disease Activity in Psoriatic Arthritis (DAPSA) | 12 weeks
  Disease Activity(DAPSA): 0-4 Remission; 5-14 Low; 15-28 Moderate; > (Greater than) 28 High Disease Activity, DAPSA = TJ (Tender Joints) + SJ (Swollen Joints) + CRP (C-reactive protein) + Activity + Pain
  1. Tender Joints Count (0-68), TJ:
  2. Swollen Joints Count (0-66), SJ:
  3. CRP (mg/dl):
  4. Patient's assessment of disease activity and pain:
  How active was your rheumatic disease on average during the last week? Scale of 1-10 (Not Active -Active)
  How would you describe the overall level of joint pain during the last week? Scale of 1-10 (None-Very Severe)

SECONDARY OUTCOMES:
Change in Psoriasis Area and Severity Index (PASI) | 24 weeks
  A measurement of the severity of psoriasis; 0 (no disease) to 72 (maximal disease)
Change in Disease Activity in Psoriatic Arthritis (DAPSA) | 24 weeks
  Disease Activity(DAPSA): 0-4 Remission; 5-14 Low; 15-28 Moderate; > (Greater than) 28 High Disease Activity DAPSA = TJ + SJ + CRP + Activity + Pain
  1. Tender Joints Count (0-68), TJ:
  2. Swollen Joints Count (0-66), SJ:
  3. CRP (mg/dl):
  4. Patient's assessment of disease activity and pain:
  How active was your rheumatic disease on average during the last week? Scale of 1-10 (Not Active -Active)
  How would you describe the overall level of joint pain during the last week? Scale of 1-10 (None-Very Severe)
Patient Reported Outcomes-Physical Function | Varying times: (at Baseline) 0,12, 24 Weeks
  -Physical Function-International Physical Activity Questionnaire (IPAQ) We will examine change in physical activity over the study (as we will be advising patients not to change exercise habits). IPAQ is an instrument for assessing levels and patterns of physical activity. IPAQ has been validated in healthy adults and is publicly available, open access, and no permissions are required for use.
Patient Reported Outcomes-Psoriatic Arthritis Disease Impact | Varying times: (at Baseline) 0, 4, 8, 12, 16, 20, 24 Weeks
  -Psoriatic Arthritis Disease Impact- Psoriatic Arthritis Impact of Disease (PSAID). The PsAID is a measure developed by the European League Against Rheumatism (EULAR) and is composed of domains selected by an international group of patients with psoriatic arthritis. The questionnaire uses a weighted scoring system (weights were derived by patient impression of importance) and has a range of 0-10 with 4 being considered a patient acceptable symptom state. The proposed Minimal Clinically Important Difference (MCID) is 3.
Patient Reported Outcomes-Skin Disease Impact | Varying times: (at Baseline) 0,12, 24 Weeks
  -Skin Disease Impact- Psoriasis Area and Severity Index (PASI). The Psoriasis Area Severity Index (PASI) is an index used to express the severity of psoriasis. It combines the severity (erythema (redness), induration (thickness) and desquamation (peeling) and percentage of affected area. This is the primary outcome measure in trials of psoriatic arthritis.
Patient Reported Outcomes-Fatigue | Varying times: (at Baseline) 0, 4, 8, 12, 16, 20, 24 Weeks
  -Fatigue- PROMIS (Patient-Reported Outcomes Measurement Information System) Fatigue (CAT) The PROMIS Fatigue scale assesses fatigue experience and impact of fatigue over 7 days. The instrument includes items on exhaustion and ability to function normally in physical, social, mental and family roles and activities. This instrument has good content validity and responsiveness in rheumatoid arthritis, a similar inflammatory arthritis. We will use the CAT (Computerized Adaptive Test) response instrument.
Patient Reported Outcomes-Depression | Varying times: (at Baseline) 0,12, 24 Weeks
  -Depression- PROMIS (Patient-Reported Outcomes Measurement Information System) Depression (CAT) The PROMIS Depression assesses sadness, guilt, self-criticism, worthlessness, loneliness, loss of interest, meaning, and purpose. The PROMIS depression scale is used across diseases but has been specifically demonstrated to have good responsiveness with therapy in patients with rheumatoid arthritis. The item bank assesses symptoms over the past 7 days. (Suicidality is not assessed in this questionnaire). We will use the CAT (Computerized Adaptive Test) response instrument.
Metabolic Profile-Blood Pressure | Varying times: (at Baseline) 0, 12, 24 Weeks
  Change in Blood Pressure Blood Pressure; BP _ systolic/diastolic; Both pressures will be assessed during the study period.
Metabolic Profile-Weight | Varying times: (at Baseline) 0, 12, 24 Weeks
  Changes in Weight; Weight_kg; Weight and Height will be combined to report BMI in kg/m^2; Body Mass Index (BMI) _ wt/h²; The standard weight status categories associated with BMI ranges for adults are listed as;
  BMI Weight Status:
  Below 18.5 Underweight 18.5 - 24.9 Normal or Healthy Weight 25.0 - 29.9 Overweight 30.0 and Above Obese
  Accessed on 11/19/19, https://www.cdc.gov/healthyweight/assessing/bmi/adult_bmi/index.html#Interpreted
Metabolic Profile-Height | Varying times: (at Baseline) 0, 12, 24 Weeks
  Height_M; Height and Weight will be combined to report BMI in kg/m^2
Metabolic Profile-Waist Measurement | Varying times: (at Baseline) 0, 12, 24 Weeks
  Waist measurement_cm
Metabolic Profile- Blood Glucose Studies | Varying times: (at Baseline) 0, 12, 24 Weeks
  Blood Glucose Studies-HbA1C; HbA1c___________ % Normal: HbA1c below 5.7% Prediabetes: HbA1c between 5.7% and 6.4 Diabetes: HbA1c of 6.5% or higher;
  Accessed on 11/19/19, https://medlineplus.gov/lab-tests/hemoglobin-a1c-hba1c-test/
Metabolic Profile- C-reactive protein | Varying times: (at Baseline) 0, 12, 24 Weeks
  C-reactive protein: General index used for inflammation
Therapy changes | Chart review at 12 and 24 Weeks
  Any changes in medications therapies will be recorded (in particular psoriatic arthritis medications, NSAIDs, cholesterol medications, high blood pressure medications, and Type 2 diabetes medications).
Preliminary Safety: Adverse event (AE)/ Serious Adverse Event (SAE) | 12 Weeks, 24 Weeks
  AEs and SAEs are reported separately. Participants can report an adverse event at any time but will be asked about it at 12 weeks and analyzed at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Ogdie-Beatty, MD, MSCE, Principal Investigator — University of Pennsylvania; Lihi Eder, MD, PhD, Principal Investigator — Women's College Hospital, University of Toronto
Locations (2):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States
- Women's College Hospital, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Manuscripts describing research results will be drafted and submitted in a timely manner for publication in widely circulated peer-reviewed journals. Physicians and researchers may request de-identified data from the PI and research plans will be reviewed on a case by case basis.